CLINICAL TRIAL: NCT02072941
Title: Preparing Spanish-speaking Older Adults for Advance Care Planning and Medical Decision Making
Brief Title: Preparing Spanish-speaking Older Adults for Advance Care Planning and Medical Decision Making (PREPARE)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: P0061026; R-1306-01500 (Other Grant/Funding Number: Patient-Centered Outcomes Research)
Record Dates: First submitted 2014-02-24; First posted 2014-02-27 (Estimated); Results first posted 2019-07-11 (Actual); Last update posted 2019-07-11 (Actual); Status verified 2019-04

CONDITIONS: Chronic Disease
Keywords: Advance care planning; Latino Health; Medical decision making; Health Literacy; Limited English proficiency; Aging
MeSH Terms: conditions — Chronic Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PREPARE intervention (Experimental): The PREPARE arm will review the PREPARE website plus the easy-to-read advance directive (AD). Participants will review PREPARE on their own for ≥20 minutes with staff present to answer questions. During PREPARE, participants answer preference questions and make an action plan (i.e., commitment to engage in advance care planning). To ensure home access to PREPARE content, participants will be given a website login and PREPARE content in digital video disc (DVD), booklet, and pamphlet format as well as the action plan and AD. One to three days before a primary care visit, the PREPARE arm will receive a reminder to come to their appointment and to bring their action plan.
  Interventions: Behavioral: PREPARE Intervention
- Control (No Intervention): The control arm will review an easy-to-read AD. Controls will review the AD for ≥15 minutes with study staff present to answer questions and will take the AD home to complete if desired. One to three days before a primary care visit, controls will receive a reminder to come to their appointment.

INTERVENTIONS:
Behavioral: PREPARE Intervention — At week 1, 3, 6, and 12 months, interviews (telephone or in person based on preference) by blinded staff will assess engagement in advance care planning (ACP), self-efficacy with ACP, and activation in and satisfaction with decision making. Blinded telephone interviews will also assess surrogate reports of patient engagement in ACP.
  Arms: PREPARE intervention

SUMMARY:
In partnership with patients, caregivers, advocacy groups and clinicians, the investigators plan to:

Aim 1: Adapt and refine PREPARE in Spanish through cognitive interviews with Spanish-speaking Latinos and stakeholders.

Aim 2: Conduct a randomized clinical trial (RCT) to compare the efficacy of PREPARE plus a previously-tested, easy-to-read- AD (intervention) versus the AD alone (control) to:

2a. Engage older Spanish-speaking Latinos in multiple ACP behaviors (i.e., identify and discuss wishes with surrogates and clinicians and complete ADs) measured by self-report, chart review, surrogate reports, and

2b. Direct observation.

2c. Improve self-efficacy and satisfaction with medical decision making.

2d. Determine whether PREPARE efficacy varies by literacy, decision control preferences, and clinician-patient language concordance.

Aim 3: Disseminate PREPARE with input from patients, surrogates, and stakeholders.

DETAILED DESCRIPTION:
PREPARE is a website (www.prepareforyourcare.org) that teaches patients how to identify what is most important in life, how to communicate their preferences to clinicians and loved ones, and how to make informed decisions. It is written at a 5th grade level and includes voice-overs of text and closed captioning of videos that model advance care planning behaviors. The goal of this proposal is to test the efficacy of PREPARE plus an easy-to-read advance directive, versus an advance directive alone, to improve patient engagement in multiple advance care planning behaviors including discussions with surrogate decision makers and clinicians in addition to advance directive completion. The investigators will also determine whether PREPARE can empower and activate patients within clinical encounters with their clinicians and help to decrease health disparities in advance care planning.

ELIGIBILITY:
Inclusion Criteria:

* Spanish-speaking adults ≥ 55 years of age
* ≥ 2 chronic illnesses determined by ICD-9 codes
* ≥ 2 visits with an outpatient primary care clinician at San Francisco General hospital in the past year
* ≥ 2 additional outpatient/inpatient visits to San Francisco General Hospital in the past year

Exclusion Criteria:

* Deaf, blind, demented or psychotic as determined by ICD-9 codes
* Too mentally or physically ill to participate as determined by their clinicians
* Moderate or severe cognitive impairment as determined by the Short Portable Mental Status Questionnaire (SPMSQ), and mild cognitive impairment by the SPMSQ plus an abnormal Mini-Cog (scores minimally affected by education/ethnicity)
* Self-reported poor vision and inability to see the words on a newspaper
* Lack of a telephone (for follow-up)
* Traveling or moving out of the area for ≥3 months during the study follow-up period.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 445 (Actual)
Dates: Start 2014-09; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Sudore, MD, Principal Investigator — University of California, San Francisco; Dean Schillinger, MD, Principal Investigator — University of California, San Francisco; Deborah E Barnes, PhD, Principal Investigator — University of California, San Francisco; John Boscardin, PhD, Principal Investigator — University of California, San Francisco; Janet Shim, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- San Francisco General Hospital and Trauma Center, San Francisco, California, United States

REFERENCES:
- [Derived] Gelfman LP, Barnes DE, Goldstein N, Volow AM, Shi Y, Li B, Sudore RL. Quality and Satisfaction With Advance Care Planning Conversations Among English- and Spanish-Speaking Older Adults. J Palliat Med. 2023 Oct;26(10):1380-1385. doi: 10.1089/jpm.2022.0565. Epub 2023 Jun 19. PMID 37335910
- [Derived] Freytag J, Street RL Jr, Barnes DE, Shi Y, Volow AM, Shim JK, Alexander SC, Sudore RL. Empowering Older Adults to Discuss Advance Care Planning During Clinical Visits: The PREPARE Randomized Trial. J Am Geriatr Soc. 2020 Jun;68(6):1210-1217. doi: 10.1111/jgs.16405. Epub 2020 Mar 10. PMID 32157684
- [Derived] Sudore RL, Schillinger D, Katen MT, Shi Y, Boscardin WJ, Osua S, Barnes DE. Engaging Diverse English- and Spanish-Speaking Older Adults in Advance Care Planning: The PREPARE Randomized Clinical Trial. JAMA Intern Med. 2018 Dec 1;178(12):1616-1625. doi: 10.1001/jamainternmed.2018.4657. PMID 30383086
- [Derived] Sudore RL, Barnes DE, Le GM, Ramos R, Osua SJ, Richardson SA, Boscardin J, Schillinger D. Improving advance care planning for English-speaking and Spanish-speaking older adults: study protocol for the PREPARE randomised controlled trial. BMJ Open. 2016 Jul 11;6(7):e011705. doi: 10.1136/bmjopen-2016-011705. PMID 27401363
- See also: PREPARE — http://www.prepareforyourcare.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study participants were enrolled from four primary care clinics associated with the San Francisco Health Network from November 2014 - March 2017. They were included if they were ≥55 years old, had ≥2 chronic medical conditions, had ≥2 visits with a PCP in the past year, and had ≥2 additional outpatient/inpatient visits in the past year.
Groups:
- PREPARE Intervention: The PREPARE arm reviewed the PREPARE website plus the easy-to-read advance directive (AD). While reviewing the PREPARE website, participants answer preference questions and make an action plan (i.e., commitment to engage in advance care planning). To ensure home access to PREPARE content, participants were given a website login and PREPARE content in digital video disc (DVD), booklet, and pamphlet format as well as the action plan and AD. One to three days before a primary care visit, participants in the PREPARE arm received a reminder phone call to come to their primary care appointment and to bring their action plan.
- Control: The control arm reviewed an easy-to-read advance directive (AD) and took the AD home to complete if desired. One to three days before a primary care visit, participants in the control arm received a reminder to come to their primary care appointment.
Period: Overall Study
Arm/Group | PREPARE Intervention | Control
Started | 219 | 226
Completed | 181 | 197
Not Completed | 38 | 29
Not completed — Withdrawal by Subject | 29 | 21
Not completed — Lost to Follow-up | 4 | 4
Not completed — Death | 3 | 2
Not completed — Removed by Study Staff | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PREPARE Intervention | Control | Total
Number analyzed (Participants) | 219 | 226 | 445
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 127 | 138 | 265
  >=65 years | 92 | 88 | 180
Age, Continuous [Mean (Standard Deviation); unit: years] | 64 (6.8) | 64 (7.2) | 64 (7.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 157 | 163 | 320
  Male | 62 | 63 | 125
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 216 | 224 | 440
  Not Hispanic or Latino | 3 | 2 | 5
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 219 | 226 | 445
Prior ACP Documentation [Count of Participants; unit: Participants] | 44 | 64 | 108

OUTCOME MEASURES:

1. Primary Outcome: New Advance Care Planning Documentation in the Medical Record at 15 Months
Description: The primary outcome is documentation of advance care planning wishes in the medical record. ACP documentation for the purposes of this study includes the easy-to-read advance directive or other valid advance directives or living wills, a durable power of attorney for healthcare document (DPOAHC), a physicians orders for life sustaining treatment (POLST) form, or other documentation of patients wishes for medical care (ie, documentation of oral directives by a physician, or code status, such as full code or do not resuscitate or do not intubate orders or notes by a physician).
Time Frame: 15 months after study enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | PREPARE Intervention | Control
Number analyzed (Participants) | 219 | 226
Participants | 83 | 58

2. Secondary Outcome: Self-reported Engagement in Advance Care Planning Behaviors
Description: Secondary outcomes were chosen to measure the full process of Advance Care Planning (ACP) using validated questionnaires, such as the patient-reported ACP Engagement Survey. This questionnaire includes both Behavior Change Process and ACP Action measures. Behavior Change Process measures include knowledge, contemplation, self-efficacy, and readiness for several ACP actions. The Process measures are assessed on an average 5-point Likert scale with a low of 1 and a high of 5, with high scores indicating more ACP engagement. Action measures include ACP actions such as identifying a surrogate decision-maker, identifying values and goals for medical care, choosing the level of leeway in surrogate decision-making, discussing one's wishes with clinicians and surrogates, and documenting one's wishes in an advance directive. Action measures use "yes" or "no" response options and are measured on a 0- to 25-point scale, where 0 is no action and 25 means they have engaged in more ACP actions.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PREPARE Intervention | Control
Number analyzed (Participants) | 219 | 226
score on a scale
  Self-reported ACP Behavior Change Process Measures | 3.2 (.07) | 2.9 (.07)
  Self-reported ACP Action Measures | 12.4 (0.53) | 10.1 (0.49)

ADVERSE EVENTS:
Time Frame: Adverse even data were collected from the day of enrollment until completion of the 12-month follow-up interview.
Arm/Group | PREPARE Intervention | Control
All-Cause Mortality (participants affected / at risk) | 3/219 | 2/226
Serious Adverse Events (participants affected / at risk) | 0/219 | 0/226
Other Adverse Events (participants affected / at risk) | 0/219 | 0/226

LIMITATIONS AND CAVEATS:
Participants could not be blinded. In addition, this study took place in one area of the country among Spanish-speaking, older patients who obtain care from safety-net settings. This may affect the generalizability of our findings.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-09-01): https://cdn.clinicaltrials.gov/large-docs/41/NCT02072941/Prot_SAP_000.pdf